CLINICAL TRIAL: NCT00537485
Title: A Placebo-controlled Study for SPM 962 in Early Parkinson's Disease Patients With Non-concomitant Treatment of L-dopa
Brief Title: A Placebo-controlled Study for SPM 962 in Early Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 243-07-001
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Early Parkinson's Disease
Keywords: SPM 962; rotigotine; Parkinson's disease; monotherapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SPM 962
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SPM 962 — transdermal application, 1 time per day
  Arms: 1
Drug: placebo — transdermal application, 1 time per day
  Arms: 2

SUMMARY:
To investigate superiority of SPM 962 over placebo in early Parkinson's disease patients in a multi-center, placebo-controlled, double-blind study following once-daily multiple transdermal doses of SPM 962 within a range of 4.5 to 36.0 mg (12-week dose titration/maintenance period)

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed as having Parkinson's disease in accordance with "Diagnostic Criteria established by the Research Committee of MHLW-specified Intractable Neurodegenerative Diseases (1995)"
2. Subject is 30 years < > 80 years at the time of informed consent
3. Hoehn & Yahr stage 1- 3
4. Total of each sum score of UPDRS Part 2 and 3 is over 10 at screening test

Exclusion Criteria:

1. Subject has previously participated in a trial with SPM 962
2. Subject is on L-dopa treatment for total of over 6 months at the time of informed consent
3. Subject has psychiatric symptoms, e.g. confusion, hallucination, delusion, excitation, delirium, abnormal behavior at screening test and baseline
4. Subject has orthostatic hypotension
5. Subject has a history of epilepsy, convulsion and other
6. Subject has a complication of serious cardiac disorder/arrhythmia or has the history
7. Subject has arrhythmia and treated with class 1a anti-arrhythmic drugs (e.g. quinidine, procainamide etc.) or class 3 anti-arrhythmic drugs (e.g. amiodarone, sotalol etc.)
8. Subject has serious ECG abnormal at screening i.e.; 1) Subject has more than 450 msec of QTc values both in two measurements at screening test 2) Subject has more than 470 msec for females and more than 450 msec for males of mean QTc values of two measurements at baseline
9. Subject has congenital long QT syndrome
10. Subject has serum potassium of less than 3.5 mEq/L at screening test.
11. Subject has total bilirubin of 3.0 mg/dL and above or AST(GOT), ALT(GPT) greater than 2.5 times (or 100 IU/L and above) of the clinical laboratory's upper limit of the reference range at screening test
12. Subject has 30 mg/dL and above of BUN or 2.0 mg/dL and above of serum creatinine at screening test
13. Subject has a history of allergy to topical medicine, e.g. transdermal patch
14. Subject is pregnant, nursing, or is child bearing potential while the trial
15. Subject is receiving therapy with prohibited drug specified in the study protocol
16. Subject has a history of pallidotomy, thalamotomy, deep brain stimulation or fetal tissue transplant
17. Subject has dementia
18. Subject is unable to give consent
19. Subject is participating in another trial of an investigational drug or done so within 12 weeks prior to the initial treatment
20. Investigator judges that subject is inappropriate as a study subject with other reasons

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — New Product Evaluation and Development
Locations (6):
- Japan (6):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- SPM962: transdermal application of SPM962, 1 time per day
- Placebo: transdermal application of placebo, 1 time per day
Period: Overall Study
Arm/Group | SPM962 | Placebo
Started | 90 | 90
Completed | 75 | 80
Not Completed | 15 | 10
Not completed — Adverse Event | 10 | 5
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Excluded 3 subjects (SPM962:2, placebo:1) because lack of assessment of efficacy, and 1 (plasebo) for not matching with the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | SPM962 | Placebo | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 35 | 71
  >=65 years | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.1) | 66.2 (7.9) | 65.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 51 | 106
  Male | 33 | 37 | 70
Region of Enrollment [Number; unit: participants]
  Japan | 88 | 88 | 176

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of Maintenance Period in Total of Each Sum Score of UPDRS Part 2 and Part 3
Description: Mean change (LOCF) from baseline to the end of maintenance period in total of each sum score of UPDRS Part 2 and Part 3.
  UPDRS is a scale for monitoring Parkinson's Disease-related disability and impairment. The UPDRS consists of the following four sub-scales. Part 1: Mentation, Part 2: Activities of Daily Living, Part 3: Motor, Part 4: Complications. Part 2 assesses 13 items and Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: baseline, end of maintenance period
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Scores on a scale | -8.4 (9.7) | -4.1 (8.2)
Statistical Analysis 1: Comparison: SPM962 vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.7 to 1.1], Standard Error of Mean 1.2

2. Secondary Outcome: Efficacy Rate in Total of Each Sum Score of UPDRS Part 2 and Part 3
Description: Effective rate (percentage of subjects with 20% or 30% decrease) (LOCF) in total of each sum score of UPDRS Part 2 and Part 3 at the end of maintenance period
Time Frame: baseline, end of maintenance period
Population: FAS, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Percentage of participants
  ≥20% decrease | 71.6 [62.2 to 81.0] | 40.9 [30.6 to 51.3]
  ≥30% decrease | 55.7 [45.3 to 66.1] | 29.5 [20.0 to 39.1]
Statistical Analysis 1: Comparison: SPM962 vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Risk Difference (RD) = 30.7, 95% CI 2-sided [16.7 to 44.6]
Statistical Analysis 2: Comparison: SPM962 vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Risk Difference (RD) = 26.1, 95% CI 2-sided [12.0 to 40.2]

3. Secondary Outcome: Mean Change in UPDRS Part 2 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score at every two weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, every two weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Week 2 | -0.6 (2.1) | -0.5 (1.3)
  Week 4 | -1.2 (2.7) | -1.0 (1.9)
  Week 6 | -1.6 (2.9) | -1.4 (2.1)
  Week 8 | -1.6 (3.3) | -1.3 (2.4)
  Week 10 | -1.7 (3.2) | -1.2 (2.7)
  Week 12 | -1.8 (3.2) | -1.1 (2.9)
  End of maintenance period | -1.8 (3.3) | -1.1 (2.9)

4. Secondary Outcome: Efficacy Rate in UPDRS Part 2 Sum Score
Description: Effective rate (percentage of subjects with 20% or 30% decrease) (LOCF) in UPDRS Part 2 sum score at every two weeks after dosing.
Time Frame: Baseline, every two weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Percentage of participants
  ≥20% decrease (Week 2) | 36.4 [26.3 to 46.4] | 13.6 [6.5 to 20.8]
  ≥20% decrease (Week 4) | 46.6 [36.2 to 57.0] | 34.1 [24.2 to 44.0]
  ≥20% decrease (Week 6) | 52.3 [41.8 to 62.7] | 40.9 [30.6 to 51.2]
  ≥20% decrease (Week 8) | 56.8 [46.5 to 67.2] | 43.2 [32.8 to 53.5]
  ≥20% decrease (Week 10) | 58.0 [47.6 to 68.3] | 38.6 [28.5 to 48.8]
  ≥20% decrease (Week 12) | 61.4 [51.2 to 71.5] | 39.8 [29.5 to 50.0]
  ≥20% decrease (End of maintenance period) | 60.2 [50.0 to 70.5] | 39.8 [29.5 to 50.0]
  ≥30% decrease (Week 2) | 20.5 [12.0 to 28.9] | 13.6 [6.5 to 20.8]
  ≥30% decrease (Week 4) | 36.4 [26.3 to 46.4] | 19.3 [11.1 to 27.6]
  ≥30% decrease (Week 6) | 43.2 [32.8 to 53.5] | 28.4 [19.0 to 37.8]
  ≥30% decrease (Week 8) | 43.2 [32.8 to 53.5] | 25.0 [16.0 to 34.0]
  ≥30% decrease (Week 10) | 43.2 [32.8 to 53.5] | 29.5 [20.0 to 39.1]
  ≥30% decrease (Week 12) | 48.9 [38.4 to 59.3] | 26.1 [17.0 to 35.3]
  ≥30% decrease (End of maintenance period) | 48.9 [38.4 to 59.3] | 26.1 [17.0 to 35.3]

5. Secondary Outcome: UPDRS Part 3 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 3 sum score at every two weeks after dosing.
  UPDRS sub-scale Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Week 2 | -2.6 (4.2) | -1.7 (3.9)
  Week 4 | -4.3 (5.2) | -2.7 (4.7)
  Week 6 | -5.7 (6.3) | -3.3 (5.3)
  Week 8 | -6.1 (6.7) | -3.3 (5.8)
  Week 10 | -6.4 (6.7) | -3.4 (5.8)
  Week 12 | -6.6 (7.2) | -3.1 (6.2)
  End of maintenance period | -6.6 (7.2) | -3.0 (6.2)

6. Secondary Outcome: Efficacy Rate in UPDRS Part 3 Sum Score
Description: as for outcome 4
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Percentage of participants
  ≥20% decrease (Week 2) | 35.2 [25.2 to 45.2] | 19.3 [11.1 to 27.6]
  ≥20% decrease (Week 4) | 52.3 [41.8 to 62.7] | 28.4 [19.0 to 37.8]
  ≥20% decrease (Week 6) | 62.5 [52.4 to 72.6] | 35.2 [25.2 to 45.2]
  ≥20% decrease (Week 8) | 67.0 [57.2 to 76.9] | 37.0 [27.4 to 47.6]
  ≥20% decrease (Week 10) | 70.5 [60.9 to 80.0] | 42.0 [31.7 to 52.4]
  ≥20% decrease (Week 12) | 70.5 [60.9 to 80.0] | 40.9 [30.6 to 51.2]
  ≥20% decrease (End of maintenance period) | 70.5 [60.9 to 80.0] | 40.9 [30.6 to 51.2]
  ≥30% decrease (Week 2) | 22.7 [14.0 to 31.5] | 15.9 [8.3 to 23.6]
  ≥30% decrease (Week 4) | 36.4 [26.3 to 46.4] | 21.6 [13.0 to 30.2]
  ≥30% decrease (Week 6) | 52.3 [41.8 to 62.7] | 23.9 [15.0 to 32.8]
  ≥30% decrease (Week 8) | 54.5 [44.1 to 64.9] | 28.4 [19.0 to 37.8]
  ≥30% decrease (Week 10) | 58.0 [47.6 to 68.3] | 29.5 [20.0 to 39.1]
  ≥30% decrease (Week 12) | 60.2 [50.0 to 70.5] | 28.4 [19.0 to 37.8]
  ≥30% decrease (End of maintenance period) | 60.2 [50.0 to 70.5] | 28.4 [19.0 to 37.8]

7. Secondary Outcome: UPDRS Part 1 Sum Score
Description: MMean change (LOCF) from baseline in UPDRS Part 1 sum score at every two weeks after dosing.
  UPDRS sub-scale Part 1 assesses 4 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Week 2 | -0.17 (0.46) | -0.01 (0.28)
  Week 4 | -0.17 (0.75) | -0.11 (0.49)
  Week 6 | -0.14 (0.89) | -0.13 (0.58)
  Week 8 | -0.23 (0.89) | -0.07 (0.56)
  Week 10 | -0.25 (0.91) | -0.11 (0.63)
  Week 12 | -0.25 (0.91) | -0.05 (0.88)
  End of maintenance period | -0.25 (0.91) | -0.05 (0.88)

8. Secondary Outcome: UPDRS Part 4 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 4 sum score at every two weeks after dosing.
  UPDRS sub-scale Part 4 assesses 11 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Week 2 | 0.19 (0.45) | 0.09 (0.33)
  Week 4 | 0.28 (0.79) | 0.08 (0.38)
  Week 6 | 0.18 (0.54) | 0.03 (0.39)
  Week 8 | 0.20 (0.61) | 0.09 (0.42)
  Week 10 | 0.19 (0.62) | 0.03 (0.44)
  Week 12 | 0.18 (0.64) | 0.05 (0.48)
  End of maintenance period | 0.18 (0.64) | 0.03 (0.47)

9. Secondary Outcome: Total of Each Sum Score of UPDRS Part 1, 2, 3, and 4
Description: Mean change (LOCF) from baseline to the end of maintenance period in total of each sum score of UPDRS Part 1, 2, 3 and 4.
  UPDRS sub-scale Part 1, 2, 3, and 4 assess 4, 13, 14, and 11 items respectively. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Week 2 | -3.3 (5.9) | -2.1 (4.6)
  Week 4 | -5.4 (7.1) | -3.8 (5.8)
  Week 6 | -7.2 (8.7) | -4.7 (6.7)
  Week 8 | -7.7 (9.4) | -4.6 (7.6)
  Week 10 | -8.1 (9.6) | -4.7 (7.7)
  Week 12 | -8.5 (9.9) | -4.1 (8.5)
  End of maintenance period | -8.5 (9.9) | -4.1 (8.5)

10. Secondary Outcome: The Modified Hoehn and Yahr Stage
Description: Mean change (LOCF) from baseline in the Modified Hoehn and Yahr Severity of Illness at the end of maintenance period. The Modified Hoehn and Yahr criteria are measured on the following 8-point scale for staging: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease without impairment of balance; 2.5, Mild bilateral disease with recovery on pull test; 3, Mild to moderate bilateral disease, some postural instability, physically independent 4, Severe disability, still able to walk or stand unassisted; and 5, Wheelchair bound or bedridden unless aided.
Time Frame: Baseline, end of maintenance period
Population: FAS, LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | SPM962 | Placebo
Number analyzed (Participants) | 86 | 88
Percentage of participants
  Increased | 8.1 | 9.1
  Not changed | 66.3 | 71.6
  Decreased | 25.6 | 19.3

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | SPM962 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/90 | 0/90
Other Adverse Events (participants affected / at risk) | 73/90 | 55/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM962 (N=90) | Placebo (N=90)
Cerebral Infarction (Vascular disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM962 (N=90) | Placebo (N=90)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Application Site Reaction (General disorders) | 42 (43) | 20 (20)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (12) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 4 (5)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hallucination (Psychiatric disorders) | 4 (5) | 0 (0)
Hallucination Visual (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 2 (2)
Nasopharyngitis (Infections and infestations) | 11 (11) | 15 (15)
Nausea (Gastrointestinal disorders) | 21 (29) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
Somnolence (Psychiatric disorders) | 13 (13) | 4 (4)
Vomiting (Gastrointestinal disorders) | 14 (22) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No